CLINICAL TRIAL: NCT04958941
Title: CUIDA-TE, an APP for the Emotional Management of the Healthcare Professionals
Brief Title: CUIDA-TE, an APP for the Emotional Management
Acronym: CUIDA-TE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UValencia_RCT_CUIDATE
Record Dates: First submitted 2021-06-09; First posted 2021-07-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Emotional Distress; Burnout, Professional; Emotional Stress
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The group will receive the ecological momentary intervention (CUIDA-TE APP). This intervention will allow the individual to learn and practice adaptive ways to regulate their emotions. The protocol contains the following components: Distraction, acceptation skills, re-appraisal and problem-solving skills.
  Interventions: Behavioral: Experimental: Intervention group
- Control group (No Intervention): This condition is a waiting list control group with no intervention. The participants will wait for a period of 3 months. They will be offered the possibility of receiving the intervention APP (CUIDA-TE) after the waiting list period.

INTERVENTIONS:
Behavioral: Experimental: Intervention group — During 2 months participants will be able to asses their mood and practice in real time their emotional regulation skills with an ecological momentary interventions APP.
  Other Names: CUIDA-TE APP
  Arms: Intervention group

SUMMARY:
The aim of this study is to develop and validate an Ecological Momentary Intervention APP for healthcare workers, in order to face of work-related stresses generated by the COVID-19 pandemic.

DETAILED DESCRIPTION:
The COVID-19 pandemic has had a very high emotional impact on healthcare workers. Ecological momentary interventions (EMI) can offer an intervention in real time, when the emotion arises. CUIDA-TE is an EMI APP based on principles of different transdiagnostic cognitive behavioral interventions focused on emotion regulation. The effectiveness of CUIDA-TE will be investigated in the current study. A two-arms randomized controlled trial (RCT) will be conducted. At least 182 healthcare workers will be randomly assigned to a 2-month immediate intervention group (CUIDA-TE APP, n= 91), or a control group (no assessment or intervention, n=91). The CUIDA-TE consists of an app-based EMI that estimates and intervenes based on ecological momentary assessment data of five emotional states: joy, fatigue, sadness, anxiety, anger, as well as sleep quality, sleep quantity, burnout, perceived stress, and self-perception of coping skills. The primary outcome is the PHQ-9. Secondary outcomes include ERQ, DERS, OASIS, BRS, SUS, and ProQOL questionnaires. Primary and secondary outcomes will be obtained at pre- and post-intervention measurements, and at 3-month follow-up measurement.

ELIGIBILITY:
Inclusion Criteria:

* to be a healthcare worker in active (from 18 until 67 years)
* to have a smartphone with Internet access and Android operating system.

Exclusion Criteria:

* to be in psychological treatment at the time of the recruitment

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Assess change in Brief Patient Health Questionnaire Mood Scale (PHQ-9) | Change from baseline(PRE), at 2 months (post intervention)and at 3 months (follow-up)
  The PHQ-9 assess depression construct and includes nine items: (1) anhedonia; (2) depressed mood; (3) trouble sleeping; (4) feeling tired; (5) change in appetite; (6) guilt, self-blame, or worthlessness; (7) trouble concentrating; (8) feeling slowed down or restless; and (9) thoughts of being better off dead or hurting oneself. PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). The PHQ-9 score is divided in the following severity categories: 5-9 (mild depression), 10-14 (modera depression), 15-19 (moderately severe depression) and 20 or greater (severe depression).
Assess change in Emotion Regulation Questionnaire (ERQ) | Change from baseline(PRE), at 2 months (post intervention)and at 3 months (follow-up)
  A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). High score indicates more likely to use this kind of emotion regulation strategies (Reappraisal Items: 1, 3, 5, 7, 8, 10; Suppression Items: 2, 4, 6, 9).
Assess change in Difficulties in Emotion Regulation Scale (DERS) | Change from baseline(PRE), at 2 months (post intervention)and at 3 months (follow-up)
  The DERS is a 36-item self-report measure of six facets of emotion regulation. Spanish validated version (Hervás & Jódar, 2008) has 28-items rated on a scale of 1 to 5. Higher scores indicate more difficulty in emotion regulation.
Assess change in Brief Resilience Scale (BRS) | Change from baseline(PRE), at 2 months (post intervention)and at 3 months (follow-up)
  The BRS is a 6-item self-report measure to assess the ability to bounce back or recover from stress. The items are rated on a 5-point scale (1 = strongly disagree; 5 = strongly agree). Range from 6 (low resilience) to 30 (high resilience).
Assess change in Burnout | Change from baseline(PRE), at 2 months (post intervention)and at 3 months (follow-up)
  Three items for assessing burnout in medical professionals. Higher score indicate more perceived burnout.
Assess change in ProQOL-V | Change from baseline(PRE), at 2 months (post intervention)and at 3 months (follow-up)
  The ProQOL (Professional Quality of Life Scale) was developed as a measure of both the negative and positive effects of working with those who have experienced traumatic stress. The ProQOL has sub-scales for compassion satisfaction, burnout, and compassion fatigue.The responses are rated on 5-point scale, indicating the frequency of each item in the last 30 days (1 = never, 2 = rarely, 3= Sometimes, 4= Often and 5 = Very Often). Higher scores on the compassion satisfaction scale represent a greater satisfaction related to the ability of the professional to be an effective caregiver in his/her job. Higher scores on the burnout scale mean a higher risk for burnout and higher scores in secondary traumatic stress indicate the professional is higher exposed to traumatic events.
Assess in usability with the System Usability Scale | At 2 months (post intervention)
  The System Usability Scale (SUS; Brooke, 1996) is a reliable, 10-item questionnaire that assess the usability of a technology application. The items are rated from 1 ("Strongly disagree") to 5 ("Strongly agree"). The scale is corrected with a formula that allows to obtain scores between 0 -100 points. Unacceptable usability (with SUS scores below 50) could indicate that a user had difficulties while using the program and could be interpreted as a barrier for the clinical effect.
Assess change in Overall Anxiety Severity and Impairment Scale (OASIS) | Change from baseline(PRE), at 2 months (post intervention)and at 3 months (follow-up)
  The OASIS is a 5-item self-report measure to assess anxiety severity and impairment

SECONDARY OUTCOMES:
Joy daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess joy/happiness daily through APP mobile. User will rate the item rating between 0 (No happiness) to 10 (Extremely happiness)
  EXAMPLE ITEM:
  Please, indicate the intensity of your CURRENT HAPPINESS 0= No happiness-------------------------------10= Extremely happy
  Item taken from mobile APP validated in Suso-Ribera C, Castilla D, Zaragozá I, Ribera-Canudas MV, Botella C, García-Palacios A. Validity, reliability, feasibility, and usefulness of pain monitor. Clin J Pain. 2018;34(10):900-8.
Fatigue daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess Fatigue daily through APP mobile. User will rate the item rating between 0 (No Fatigue) to 10 (Extreme fatigue)
  EXAMPLE ITEM:
  Please, indicate the intensity of your CURRENT FATIGUE 0= No fatigue--------------------------------10= Extreme fatigue
  Item taken from mobile APP validated in Suso-Ribera C, Castilla D, Zaragozá I, Ribera-Canudas MV, Botella C, García-Palacios A. Validity, reliability, feasibility, and usefulness of pain monitor. Clin J Pain. 2018;34(10):900-8.00-8.
Sadness daily item integrated in the APP mobile | During intervention process up to 2 months
  Item from mobile APP validated in Suso-Ribera C, Castilla D, Zaragozá I, Ribera-Canudas MV, Botella C, García-Palacios A. Validity, reliability, feasibility, and usefulness of pain monitor. Clin J Pain. 2018;34(10):900-8.
Anxiety daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess Anxiety daily through APP mobile. User will rate the item rating between 0 (No Anxiety) to 10 (Extremely Anxious)
  EXAMPLE ITEM:
  Please, indicate the intensity of your CURRENT ANXIETY 0= No anxiety-----------------------------10= Extremely anxious
  Item taken from mobile APP validated in Suso-Ribera C, Castilla D, Zaragozá I, Ribera-Canudas MV, Botella C, García-Palacios A. Validity, reliability, feasibility, and usefulness of pain monitor. Clin J Pain. 2018;34(10):900-8.
  Item from mobile APP validated in Suso-Ribera C, Castilla D, Zaragozá I, Ribera-Canudas MV, Botella C, García-Palacios A. Validity, reliability, feasibility, and usefulness of pain monitor. Clin J Pain. 2018;34(10):900-8.
anger daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess Anger daily through APP mobile. User will rate the item rating between 0 (No Anger) to 10 (Extremely Angry)
  EXAMPLE ITEM:
  Please, indicate the intensity of your CURRENT ANGER 0= No anger-------------------------------10= Extremely angry
  Item from mobile APP validated in Suso-Ribera C, Castilla D, Zaragozá I, Ribera-Canudas MV, Botella C, García-Palacios A. Validity, reliability, feasibility, and usefulness of pain monitor. Clin J Pain. 2018;34(10):900-8.
sleep quality daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess sleep quanlity daily through APP mobile. User will rate if the work have interfered with the quality of sleep rating between 0 (No interference) to 10 (maximum interference)
  EXAMPLE ITEM:
  Has WORK interfered with the quality of your SLEEP tonight? 0 = No Interference----------------------10 = Maximum Interference
  Item elaborated AD HOC for this study
sleep quantity daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess sleep quantity daily through APP mobile. The user will rate the number of hours of sleep each day.
  EXAMPLE ITEM:
  How many hours have you slept in the last 24 hours?
  Item elaborated AD HOC for this study
burnout daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess the degree of perceived burnout daily through APP mobile. User will rate the item rating between 0 (Totally disagree) to 10 (Totally agree)
  EXAMPLE ITEM:
  Please, indicate your degree of agreement with the next statement: "I am burned out from my work" 0= totally disagree----------------------------------------10= totally agree
  Item adapted from West CP, Dyrbye LN, Sloan JA, Shanafelt TD. Single item measures of emotional exhaustion and depersonalization are useful for assessing burnout in medical professionals. JGen Intern Med. 2009; 24(12):1318-1321. https://doi.org/10.1007/s11606-009-1129-z PMID: 19802645
perceived stress daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess perceived stress daily through APP mobile. User will rate the item rating between 0 (No stress) to 10 (Extremely stressed)
  EXAMPLE ITEM:
  Please, indicate the intensity of your CURRENT STRESS 0= No stress------------------------------10= Extremely stressed
  Item created AD HOC for this study.
self-perception of coping skills daily item integrated in the APP mobile | During intervention process up to 2 months
  Item to assess perceived self-perception of coping skills daily through APP mobile.
  User will rate the item rating between 0 (No capable) to 10 (Extremely capable)
  EXAMPLE ITEM:
  To what extent do you feel CAPABLE OF COPING with your problems right now? 0= No capable---------------------------------10= Extremely capable
  Item created AD HOC for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Castilla, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castilla D, Navarro-Haro MV, Suso-Ribera C, Diaz-Garcia A, Zaragoza I, Garcia-Palacios A. Ecological momentary intervention to enhance emotion regulation in healthcare workers via smartphone: a randomized controlled trial protocol. BMC Psychiatry. 2022 Mar 5;22(1):164. doi: 10.1186/s12888-022-03800-x. PMID 35248015
- See also: CUIDA-TE APP — http://emi.labpsitec.es/